CLINICAL TRIAL: NCT02722642
Title: A Single-center, Non-randomized, Before-and-after Self Control Study of Bronchial Basal Cell Transplantation for Bronchiectasis Treatment
Brief Title: Autologous Bronchial Basal Cells Transplantation for Treatment of Bronchiectasis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regend Therapeutics (Industry)
Collaborators: Southwest Hospital, China (Other); Tongji University (Other)
Responsible Party: Principal Investigator, Xiaotian Dai, Principal Investigator, Regend Therapeutics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201602301
Record Dates: First submitted 2016-03-09; First posted 2016-03-30 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchial basal cells (Experimental): Patients will receive 10^6 (1 million)/Kg/person cells of clinical grade bronchial basal cells (BBCs) injected via fiberoptic bronchoscopy after fully lavage of the localized lesions.
  Interventions: Biological: Bronchial basal cells

INTERVENTIONS:
Biological: Bronchial basal cells — Patients will receive 10^6 (1 million) /Kg/person cells of clinical grade bronchial basal cells (BBCs) injected via fiberoptic bronchoscopy after fully lavage of the localized lesions.

SUMMARY:
Bronchiectasis is a result of chronic inflammation compounded by an inability to clear mucoid secretions. Inflammation results in progressive destruction of the normal lung architecture, in particular the elastic fibers of bronchi. Currently there is no effective drug for bronchiectasis. This study intends to carry out an open, single-center, non-randomized, self control phase I/II clinical trial. During the treatment, bronchial basal cells (BCCs) will be isolated from patients' own bronchi by bronchoscopic brushing and expanded in vitro. Cultured cells will be injected directly into the lesion by fiberoptic bronchoscopy after lavage. After six-month observation, the investigators will evaluate the safety and effectiveness of the treatment by measuring the key indicator-- the CT imaging of dilated bronchi as well as four secondary indicators including the pulmonary function, laboratory factor level, incidence of acute exacerbation and the patients' self-evaluation.

DETAILED DESCRIPTION:
Bronchiectasis is a term for irreversible lung damage resulting from recurrent episodes of infection and inflammation. Bronchial basal cells (BCCs) have been proven with stem cell activity to regenerate bronchi and repair lung damage. In this single-center, non-randomized, self control phase I/II clinical trial, patients' own BCCs will be grown in laboratory before injected to the damaged part of lung tissue. Transplanted BCCs have the potential to replenish the bronchial epithelium and reconstruct respiratory architecture.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed as bronchiectasis.
* Subjects with at least 6 lung segments affected.
* Subjects with stable condition for more than 2 weeks.
* Subjects can tolerate bronchoscopy.
* Subjects signed informed consent.

Exclusion Criteria:

* Women of childbearing age at the stage of pregnancy or lactation, or those without taking effective contraceptive measures.
* Subjects with syphilis or HIV positive antibody.
* Subjects with any malignancy.
* Subjects suffering from any of the following pulmonary diseases: active tuberculosis, pulmonary embolism, pneumothorax, multiple huge bullae, uncontrolled asthma, acute exacerbation of chronic bronchitis or extremely severe COPD.
* Subjects suffering from other serious diseases, such as diabetes, myocardial infarction, unstable angina, cirrhosis, and acute glomerulonephritis.
* Subjects with leukopenia (WBC less than 4x10^9 / L) or agranulocytosis (WBC less than 1.5x10^9 / L or neutrophils less than 0.5x10^9 / L) caused by any reason.
* Subjects with severe renal impairment, serum creatinine> 1.5 times the upper limit of normal.
* Subjects with liver disease or liver damage: ALT, AST, total bilirubin> 2 times the upper limit of normal.
* Subjects with a history of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
* Subjects with severe arrhythmias (such as ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter, etc.) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
* Subjects with a history of alcohol or illicit drug abuse.
* Subjects accepted by any other clinical trials within 3 months before the enrollment.
* Subjects with poor compliance, difficult to complete the study.
* Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
CT imaging of dilated bronchi | 3 day - 6 months
  CT image of dilated bronchi will be analyzed.Clinical indicators include the spread of dilation, extent of dilation and the thickness of bronchi wall.

SECONDARY OUTCOMES:
6-minute walk distance test | 3 day - 6 months
MRC chronic dyspnea scale | 3 day - 6 months
St. George's Respiratory Questionnaire (SGRQ) scale | 3 day - 6 months
inflammation indicators | 3 day - 6 months
  TNF-α,IL1-β,PDGF,MMP9,TIMP1,CRP, PCT
fibrotic factor level | 3 day - 6 months
  TGF-β, Hydroxyproline
incidence of acute exacerbation | 3 day-6 months
patients' self-evaluation | 3 day - 6 months
  The self-efficacy evaluation can also be classified into four levels: effective, improved, stable and invalid.
blood gas level（PH） | 3 day - 6 months
blood gas level（HCO3） | 3 day - 6 months
blood gas level（PaCO2） | 3 day - 6 months
blood gas level（PaO2） | 3 day - 6 months
pulmonary function test (DLco) | 3 day - 6 months
  Diffusing capacity of CO
pulmonary function test (FEV1) | 3 day - 6 months
  Forced expiratory volume in one second, FEV1
pulmonary function test (FVC) | 3 day - 6 months
  forced vital capacity
pulmonary function test (MVV) | 3 day - 6 months
  maximal voluntary ventilation
pulmonary function test (MMEF) | 3 day - 6 months
  maximal midexpiratory flow curve

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zuo, Ph.D., Study Chair — Regend Therapeutics Co.Ltd
Locations (1):
- First Affiliated Hospital of the Third Military University, PLA (Southwest Hospital), Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuo W, Zhang T, Wu DZ, Guan SP, Liew AA, Yamamoto Y, Wang X, Lim SJ, Vincent M, Lessard M, Crum CP, Xian W, McKeon F. p63(+)Krt5(+) distal airway stem cells are essential for lung regeneration. Nature. 2015 Jan 29;517(7536):616-20. doi: 10.1038/nature13903. Epub 2014 Nov 12. PMID 25383540